CLINICAL TRIAL: NCT03626584
Title: Molecular Imaging in Cardiovascular Disease Using Hybrid Positron Emission Tomography/Magnetic Resonance Imaging (PET/MR): Cardiac Amyloidosis
Brief Title: PET/MR Imaging In Patients With Cardiac Amyloidosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC17011
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac Amyloidosis Patients: Patients with established diagnosis of cardiac amyloidosis.
  Interventions: Other: 18F-NaF PET
- Healthy Volunteers: Healthy volunteer subjects of similar age and gender to patient cohort.
  Interventions: Other: 18F-NaF PET

INTERVENTIONS:
Other: 18F-NaF PET — Hybrid 18F-NaF PET/MR imaging for observational diagnostic purposes

SUMMARY:
PET scanning (positron emission tomography) is a well-established technique used to identify areas of interest within the body. It involves injecting a radioactive tracer which highlights abnormal areas. It has recently been combined with CT (computed tomography) and MRI (magnetic resonance imaging) scanning to more accurately identify abnormalities within the heart. Cardiac amyloidosis, a condition which causes thickening of heart muscle due to abnormal protein deposits, is of particular interest. There are different forms of this condition and at present samples of tissue need to be taken and analysed in order to assess these accurately, which carries risks.

The study makes use of hybrid PET/MR scanning using a designated scanner which enables PET scanning combined with MRI scanning. The investigators will use a PET tracer which is widely used in cardiac imaging as it is hoped this will enable characterisation of abnormal areas within the heart in this condition in a way which hasn't been done before.

All participants will undergo PET scanning, where a radioactive tracer is injected into a vein before the scan. The radioactive substance only lasts for a short time and is safe, passed out of the body in urine. If successful, this imaging method will enable us to detect differences between different forms of cardiac amyloidosis in a non-invasive way, improving the diagnostic capabilities in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 40 years
* Completion of informed consent
* Established diagnosis of cardiac amyloidosis

Exclusion Criteria:

* Inability or unwilling to give informed consent
* Women who are pregnant, breastfeeding or of child-bearing potential (women who have experienced menarche, are pre-menopausal and have not been sterilised) will not be enrolled into the trial.
* Major intercurrent illness with life-expectancy <2 years.
* Renal dysfunction (eGFR less than or equal to 30ml/min/1.73m2)
* Adverse reaction or hypersensitivity to 18F-FDG PET tracer
* NYHA Class IV heart failure
* Patients with atrial fibrillation and poor rate control
* Contraindications to MRI scanning
* Previous history of contrast allergy of adverse reactions (Gadolinium-containing agents)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the Edinburgh Heart Centre will be invited to participate. Inpatients and outpatients are eligible. Healthy volunteers will be invited to participate by local recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Myocardial 18F-NaF uptake | 1 year
  Quantification of myocardial PET tracer uptake

CONTACTS AND LOCATIONS:
Overall Officials: Marc R Dweck, MD PhD, Study Director — University of Edinburgh
Locations (1):
- Queen's Medical Research Institute, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No